CLINICAL TRIAL: NCT02758899
Title: The Effects of Diabetes and Glycosylation Profile on Outcomes in the Surgical Treatment of Cervical Spondylosis
Brief Title: Diabetes and Glycosylation in Cervical Spondylosis
Status: Terminated | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201309048
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Diabetes; Cervical Myelopathy; Cervical Spondylosis
Keywords: Anterior cervical discectomy; Anterior cervical fusion
MeSH Terms: conditions — Diabetes Mellitus; Spondylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetic Patients: Patients with diagnosis of type I or type II diabetes, in addition to clinical diagnosis of cervical myelopathy or cervical spondylosis requiring anterior cervical discectomy and fusion.
- Control Patients: Patients with no diagnosis of diabetes, with a clinical diagnosis of cervical myelopathy or cervical spondylosis requiring anterior cervical discectomy and fusion.

SUMMARY:
The purpose of this study is to determine the relevant significance of diabetes on cervical disc degeneration, and correlate diabetic control (HgbA1C) with disc glycosylation profile in patients undergoing anterior cervical discectomy and fusion for cervical spondylosis. Additionally, to compare the level of degenerative cervical disc glycosylation in patients with and without diabetes.

Hypothesis: Patients with diabetes and degenerative cervical disc disease have higher levels of disc tissue glycosylation, and higher levels of glycosylation are correlated with poor outcomes.

DETAILED DESCRIPTION:
Spine surgery has increased substantially in the U.S. during the past decade, with an estimated 100,000 patients undergoing cervical procedures annually. As the demographics of an aging population begin to increase their utilization of healthcare resources, surgeons will undoubtedly be faced with an increasing number of high-risk patients. A number of factors including smoking, obesity, and diabetes significantly contribute to surgical complications following spinal arthrodesis. Nicotine has a direct inhibitory effect on autologous cancellous bone graft revascularization, significantly increasing the rate of bony non-union. Similarly, obesity has been demonstrated to represent a significant risk factor for subsequent pseudoarthrosis and has been linked to nearly a 100% higher in-hospital complication rate. Spine instrumentation in the setting of diabetes has been linked to reduced incidence of bony fusion, increased surgical site infection9, and higher hospital costs.

Achieving solid bony fusion following cervical arthrodesis has long been considered the most important primary outcome measure and is highly correlated with patient reported outcome measures. Non-union or pseudoarthrosis following cervical instrumentation can lead to persistent neck pain and/or recurrence of myeloradiculopathy. The incidence of bony fusion is affected by both patient systemic factors and local biologic environment. Significant resources have been invested into studying local environment following spinal arthrodesis, with a particular focus on high-risk patients. Animal studies have suggested diabetes is a significant risk factor for disc degeneration, yet corresponding human studies are lacking. Understanding the mechanism by which diabetes contributes to disc degeneration is the first requisite step in designing therapies to prevent diabetes associated disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* A diagnosis of type I or type II diabetes mellitus (diabetes cohort only)
* Clinical diagnosis of cervical myelopathy or cervical spondylosis
* Requiring anterior cervical discectomy and fusion
* Able to cooperate in the completion of standardized outcome measures (NDI)
* Willing and able to comply with study protocol
* Control patients will fulfill all eligibility criteria with the exception of diagnosis of diabetes.

Exclusion Criteria:

* Pre-existent neurologic disorder or mental disorder that would preclude accurate evaluation (psychiatric disease, Parkinson's disease, Alzheimer's disease)
* History of previous anterior cervical fusion adjacent to the operative site
* Osteoporosis
* Rheumatoid arthritis
* Pregnancy
* Active malignancy
* History of previous posterior cervical decompression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical diagnosis of cervical myelopathy or cervical spondylosis that require an anterior cervical discectomy and fusion.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Z Ray, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diabetic Patients | Control Patients
Started | 11 | 10
Completed | 9 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: There were 11 diabetic patients consented, but 2 were withdrawn. One declined surgery and the other, we could not collect sample due to emergent surgery. Therefore, we have results on 9 diabetic pts. Controls - we started with 10. No sample was collected on one subject, so we ended with 9. This explains difference in participant flow numbers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetic Patients | Control Patients | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 7 | 2 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Absolute Disc Glycosylation Levels
Description: After extraction during surgery, the intervertebral disc will be sent in saline to the lab for glycosylation analysis. Glycosylation refers to the chemical bonds of blood glucose to the red blood cells. Normally, only a small percentage of blood glucose, usually between 4.5%- 6%, is covalently linked to the red blood cells in hemoglobin of the non diabetes population.
Time Frame: One-time, measured at time of surgery
Measure: Number; unit: R2 of glycosylation in the disc
Arm/Group | Diabetic Patients | Control Patients
Number analyzed (Participants) | 9 | 9
R2 of glycosylation in the disc | 0.0528 | 0.44065

2. Secondary Outcome: Neck Disability Index (NDI)
Description: Questionnaire to determine how subject's neck pain has affected their ability to manage in everyday life. Scores are calculated. Low scores indicate less pain/less disability. High scores indicate more pain/more disability. Scores range from 0-100.
Time Frame: 24 months
Population: Neck Disability Index questionnaires were given to all patients in the study pre-operatively and at set intervals post-operatively. The study ended earlier than originally anticipated. The number of questionnaires that were completed were not enough to do a thorough analysis.
Arm/Group | Diabetic Patients | Control Patients
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rates of Fusion
Description: Rate of fusion will be assessed by flexion extension X-rays at routine follow-up, translation method (<2mm) and/or by computed tomography (CT) scan at 2 year post- operatively.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 2 years after surgery.
Arm/Group | Diabetic Patients | Control Patients
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No